CLINICAL TRIAL: NCT05364203
Title: Interest of Immersive Virtual Reality on Stress During Botulinum Toxin Injections in Spasticity
Brief Title: Interest of Immersive Virtual Reality on Stress During Botulinum Toxin Injections in Spasticity (RVTOX)
Acronym: RVTOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: RBHP 2021 PLAN PAQUET; 2021-A02631-40 (Other: ANSM)
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-10

CONDITIONS: Central Neurogical Impairment
Keywords: central neurological impairment (stroke, multiple sclerosis); virtual reality mask; spasticity; botulinum toxin injections; stress; pain
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Muscle Spasticity; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be selected during the physical medicine and rehabilitation consultation of the MPR department. They will be given the protocol newsletter. After their agreement to participate in the study, the following data will then be collected: age, sex, pathology, date of the first botulinum toxin injection. Randomization can then take place. The injections will be performed in day hospitalization. During the 1st injection, no particular device will be used. The following injections will be performed with the mask off or with virtual reality will be the randomization scheme.
  The stress before, during and after the 1st and the last injection will be measured at each session by collecting the frequency variability by a heart rate monitor or equivalent, in four stages, at rest, before the procedure, during the procedure and after the procedure), during the 1st and last injection at each session. Pain during injection will be assessed using a vertical visual analogue scale.
Who Masked: Investigator
Masking Description: The processing of the heart rate data will be carried out blind from the device used. Indeed, the investigator must not be aware of the device used during the session so as not to have an influence and draw hasty conclusions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- no intervention (No Intervention): Injections were done as usual without mask.
- Comparator (Active Comparator): Injections are made as in standard practice. The virtual reality headset is added to the patient. In this case, there is no image or sound. The mask is off.
  Interventions: Device: DEEPSEN virtual reality mask
- Intervention (Experimental): Injections are made as in standard practice. We add the virtual reality mask with the image and the sound.
  Interventions: Device: DEEPSEN virtual reality mask

INTERVENTIONS:
Device: DEEPSEN virtual reality mask — DEEPSEN virtual reality mask with 360 ° vision. The audio-visual content will be chosen by the patient.
  Arms: Comparator; Intervention

SUMMARY:
The main objective of the study is to investigate the effect of exposure to a virtual reality session during botulinum toxin injections on injection-induced stress.

The secondary objectives are to study the effect of exposure to a virtual reality session during botulinum toxin injections, on the pain induced by the injection. And study the evolution of the effects of virtual reality with the repetition of the sessions.

DETAILED DESCRIPTION:
Botulinum toxin injections is very frequently used in the treatment of spasticity after central neurological damage (stroke, multiple sclerosis, spinal cord injury, head trauma). The injections may be painful and the tolerance of the injections varies from one patient to another. The pain felt during the injection causes in most patients great stress during the injection.

Virtual reality is a video technique with 360 ° vision simulating the physical presence of the patient in an "existing" environment outside the hospital setting. This technique has been used in painful procedures but only one publication, in pediatrics, has shown a decrease in pain and agitation during botulinum toxin injections.

The hypothesis of this research is that an immersive virtual reality system can, in adults, reduce stress and the painful experience of botulinum toxin injections.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, suffering from spasticity of neurological origin (multiple sclerosis, stroke, head trauma, etc.) and eligible for treatment by botulinum toxin injection
* Able to give an informed consent to participate in research
* Affiliation to Social Security.

Exclusion Criteria:

* Contraindication to virtual reality (epilepsy, schizophrenia, strabismus, amblyopia, anisometropia, local contraindication to wearing a helmet (lesion of the face or the skull)
* Major cognitive disorders
* Any medical condition deemed by the investigator to be incompatible with the research.
* Indication of sedation by MEOPA during botulinum toxin injection sessions.
* Patients who have already experienced virtual reality
* Drug treatment or medical condition that may affect heart rate variability
* Pregnant or breastfeeding women
* Patients under safeguard of justice
* Refusal of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) before injection and during the injections | during the procedure
  The stress measurement is carried out using a watch and a belt (heart rate monitor) which, thanks to several parameters, will allow us to carry out an HRV analysis on the KUBIOS software.

SECONDARY OUTCOMES:
Effect on the pain induced by the injection | during the procedure
  At the end of the injections, the doctor asks the patient to give a score between 0 (no pain) and 10 (the worst pain), in order to give an idea of the pain felt during the botulinum toxin injections.
Quality of the conditions for performing botulinum toxin injections | during the procedure
  Estimate by the doctor immediately after the end of the session [by a simple numerical scale (ENS) ranging from 0 ("extremely bad conditions") to 10 ("extremely good conditions")] or [on a 5-point Likert type scale points (conditions extremely bad/poor/neither bad nor good/good/extremely good)]

CONTACTS AND LOCATIONS:
Overall Officials: Lech DOBIJA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France, France

IPD SHARING:
Plan to Share IPD: Yes
According to the provisions concerning data confidentiality that are available to those responsible for the quality control of biomedical research, all researchers with direct access to the data will take the necessary precautions to ensure the confidentiality of information (participant identification and results). All data collected will be anonymized. Our study will be continued by the investigator and a second article with the results will be published. Dissemination of the results of this study will be through peer-reviewed publications, and national and international conferences

REFERENCES:
- [Derived] Bougeard M, Hauret I, Pelletier-Visa M, Plan-Paquet A, Givron P, Badin M, Pereira B, Lanhers C, Coudeyre E. Use of immersive virtual reality for stress reduction during botulinum toxin injection for spasticity (RVTOX): a study protocol of a randomised control trial. BMJ Open. 2023 Oct 30;13(10):e066726. doi: 10.1136/bmjopen-2022-066726. PMID 37903608